CLINICAL TRIAL: NCT06260826
Title: Comparison of Continuous Positive Airway Pressure Modes (Constant Via Facial Mask vs. Auto Via Nasal Mask) on Oxygenation and Pulmonary Function in Elderly Patients After Major Open Abdominal Surgery
Brief Title: CPAP on Oxygenation and Pulmonary Function in Elderly Patients After Major Open Abdominal Surgery
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Dang Thu (Other)
Responsible Party: Sponsor-Investigator, Nguyen Dang Thu, Principal Investigator, Vietnam Military Medical University
Organization: Vietnam Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3977/QĐ-HVQY
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Continuous Positive Airway Pressure; Pulmonary Function; Older People
Keywords: Continuous Positive Airway Pressure; Pulmonary Function; Elderly patients; Abdominal open surgery

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned in a 1:1 ratio to either the O2-Max Trio or JPAP group through a computer-generated randomization list .
Masking Description: the treatment allocation was unblinded to both the patient and the staffs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Auto-CPAP via nasal mask (Experimental): Patients connected to the JPAP system (Metran, Saitama, Japan) via a nasal mask with the initial CPAP 2 cmH2O, then reach CPAP 7.5 cmH2O after a ramping time of 5 minutes.
  Interventions: Device: Auto CPAP via nasal mask (JPAP machine)
- Constant-CPAP via facial mask (Active Comparator): Patients connected to the O2-Max Trio CPAP system (Pulmodyne, Indianapolis, USA) with a facial mask and maintained a CPAP at 7.5 cm H2O
  Interventions: Device: Constant CPAP via facial mask (O2-Max Trio system)

INTERVENTIONS:
Device: Auto CPAP via nasal mask (JPAP machine) — Auto Continuous Positive Airway Pressure via nasal mask using the JPAP system (Metran, Saitama, Japan) which can provide CPAP with a range of 2-10 cmH2O, the initial CPAP 2 cmH2O, then reach 7.5 cmH2O after a ramping time. CPAP values may vary with each breath until the obstruction is resolved
  Arms: Auto-CPAP via nasal mask
Device: Constant CPAP via facial mask (O2-Max Trio system) — Patients connected to the O2-Max Trio CPAP system (Pulmodyne, Indianapolis, USA) with a facial mask that was adjusted to maintain a CPAP at 7.5 cm H2O and FiO2 30% continuously for the following 1 hour
  Arms: Constant-CPAP via facial mask

SUMMARY:
Postoperative continuous positive airway pressure (CPAP) can improve lung function. The risk of pulmonary complications is high after major abdominal surgery but may be reduced by prophylactic postoperative noninvasive ventilation using CPAP. This study compared the effects of auto-CPAP via a nasal mask (JPAP) and constant-CPAP via a facial mask (O2-Max Trio) on oxygenation and pulmonary function in elderly patients after major open abdominal surgery.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo screening period to determine eligibility for study entry.

Patients aged over 60 years, scheduled for major open abdominal surgery (i.e., gastrectomy, colectomy, proctocolectomy, or abdominal aortic aneurysm repair).

All patients received standardized anesthetic management following the established protocols of our hospital. Before induction, an epidural catheter was placed in the epidural space at thoracic T7-9 level for upper abdominal surgery and at lumbaric L1-3 level for lower abdominal surgery. A 0.2% bupivacaine solution was administered with a 5 ml bolus dosage, maintained at 5 ml/h during surgery, and the infusion rate was adjusted for pain management until postoperative day 3. General anesthesia was induced using propofol, fentanyl, and rocuronium, with maintenance using sevoflurane. Neuromuscular blockade was monitored using the train-of-four (TOF) stimulation. Fentanyl and epidural infusion rates were adjusted to maintain the Surgical Pleth Index (SPI) in the range of 40-70. Extubation was only performed when the TOF ratio was > 90%.

In the PACU, after extubation, all patients lay on their backs with a backrest tilted to 45 degrees. Postoperative pain was assessed using a numeric rating scale (NRS; 0-10) and treated with epidural boluses or IV opioids if pain exceeded NRS 3 at rest or NRS 5 during movement. Acute pain, nausea, or circulatory problems were managed and ruled out. CPAP was administered when patients were conscious and had the ability to cough and expectorate phlegm.

Patients were randomly assigned in a 1:1 ratio to either the O2-Max Trio or JPAP group through a computer-generated randomization list.

Patients in the O2-Max Trio group received CPAP via the O2-Max Trio CPAP system (Pulmodyne, Indianapolis, USA) with a facial mask that was adjusted to maintain a CPAP at 7.5 cm H2O and FiO2 30% continuously for the following 1 h.

JPAP group patients connected to the JPAP system (Metran, Saitama, Japan) via a nasal mask with the initial CPAP 2 cmH2O, then reach CPAP 7.5 cmH2O after a ramping time of 5 minutes.

Discharge from the PACU was according to a modified Aldrete discharge score. The criteria for discharge from the PACU were hemodynamic stability, SpO2 .90% with FIO2,0.4, absence of clinical signs of respiratory distress, full consciousness, and sufficient diuresis (>0.3 ml/kg/h).

ELIGIBILITY:
Inclusion Criteria:

* Patient agrees to participate in the study
* Age 60 or older
* ASA I, II, III
* Patients underwent open abdominal surgery under general anesthesia, and extubation without complications

Exclusion Criteria:

* Upper airway deformities
* Significant bullous emphysema
* Bronchopleural fistula
* Facial deformation
* Non-epidural anesthesia
* Hemodynamic unstable
* Inability to provide consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The oxygenation-PaO2/FiO2 | Three time points: Before surgery, arrival at the post-anesthesia care unit (before CPAP), and 1 hour after CPAP
  The partial pressure of oxygen in arterial blood (PaO2)/fraction of inspired oxygen (FIO2) ratio. PaO2 was measured by drawing 2 mL of blood from the radial artery and using a Cobas B221 blood gas analyzer (Roche, Basel, Switzerland), whereas the FIO2 was read from the CPAP apparatus.

SECONDARY OUTCOMES:
The forced vital capacity (FVC) | Three time points: Before surgery, arrival at the post-anesthesia care unit (before CPAP), and 1 hour after CPAP
  Forced vital capacity (FVC) was evaluated by spirometry test. The parameter was measured with Spirobank II Advanced (Medical International Research, Roma, Italia)
The forced expiratory volume in the first second-FEV1 | Three time points: Before surgery, arrival at the post-anesthesia care unit (before CPAP), and 1 hour after CPAP
  The forced expiratory volume in the first second-FEV1 was evaluated by spirometry test.
  The parameter was measured with Spirobank II Advanced (Medical International Research, Roma, Italia)
The FEV1/FVC ratio | Three time points: Before surgery, arrival at the post-anesthesia care unit (before CPAP), and 1 hour after CPAP
  The FEV1/FVC ratio was evaluated by spirometry test. The parameter was measured with Spirobank II Advanced (Medical International Research, Roma, Italia)
The peak expiratory flow-PEF | Three time points: Before surgery, arrival at the post-anesthesia care unit (before CPAP), and 1 hour after CPAP
  The peak expiratory flow-PEF was evaluated by spirometry test. The parameter was measured with Spirobank II Advanced (Medical International Research, Roma, Italia)

CONTACTS AND LOCATIONS:
Overall Officials: Thu Nguyen Dang, Principal Investigator — Vietnam Military Medical University
Locations (1):
- VietXo Friendship Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osterkamp JTF, Strandby RB, Henningsen L, Marcussen KV, Thomsen T, Mortensen CR, Achiam MP, Jans O. Comparing the effects of continuous positive airway pressure via mask or helmet interface on oxygenation and pulmonary complications after major abdominal surgery: a randomized trial. J Clin Monit Comput. 2023 Feb;37(1):63-70. doi: 10.1007/s10877-022-00857-7. Epub 2022 Apr 16. PMID 35429325
- [Background] Garutti I, Puente-Maestu L, Laso J, Sevilla R, Ferrando A, Frias I, Reyes A, Ojeda E, Gonzalez-Aragoneses F. Comparison of gas exchange after lung resection with a Boussignac CPAP or Venturi mask. Br J Anaesth. 2014 May;112(5):929-35. doi: 10.1093/bja/aet477. Epub 2014 Feb 3. PMID 24496783
- [Background] Ireland CJ, Chapman TM, Mathew SF, Herbison GP, Zacharias M. Continuous positive airway pressure (CPAP) during the postoperative period for prevention of postoperative morbidity and mortality following major abdominal surgery. Cochrane Database Syst Rev. 2014 Aug 1;2014(8):CD008930. doi: 10.1002/14651858.CD008930.pub2. PMID 25081420
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Abbott TEF, Fowler AJ, Pelosi P, Gama de Abreu M, Moller AM, Canet J, Creagh-Brown B, Mythen M, Gin T, Lalu MM, Futier E, Grocott MP, Schultz MJ, Pearse RM; StEP-COMPAC Group. A systematic review and consensus definitions for standardised end-points in perioperative medicine: pulmonary complications. Br J Anaesth. 2018 May;120(5):1066-1079. doi: 10.1016/j.bja.2018.02.007. Epub 2018 Mar 27. PMID 29661384
- [Background] Ferreyra GP, Baussano I, Squadrone V, Richiardi L, Marchiaro G, Del Sorbo L, Mascia L, Merletti F, Ranieri VM. Continuous positive airway pressure for treatment of respiratory complications after abdominal surgery: a systematic review and meta-analysis. Ann Surg. 2008 Apr;247(4):617-26. doi: 10.1097/SLA.0b013e3181675829. PMID 18362624
- [Background] Hulzebos E. Continuous positive airway pressure reduces respiratory complications following abdominal surgery. Aust J Physiother. 2008;54(3):217. doi: 10.1016/s0004-9514(08)70031-x. No abstract available. PMID 18833685